CLINICAL TRIAL: NCT00939952
Title: Ertapenem Pharmacokinetics in Patients in Continuous Ambulatory Peritoneal Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany College of Pharmacy and Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Katie Cardone, Assistant Professor, Albany College of Pharmacy and Health Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 35922; 09-006
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-01

CONDITIONS: Continuous Ambulatory Peritoneal Dialysis; End Stage Renal Disease
Keywords: ertapenem; CAPD; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ertapenem 500 mg IV x1 (Active Comparator): All patients will receive ertapenem 500 mg IV once.
  Interventions: Drug: ertapenem

INTERVENTIONS:
Drug: ertapenem — 500 mg IV once
  Other Names: Invanz

SUMMARY:
The objective of this study is to characterize the pharmacokinetic profile of ertapenem during continuous ambulatory peritoneal dialysis (CAPD).

DETAILED DESCRIPTION:
BACKGROUND:

Infection is a leading cause of morbidity and mortality in end-stage renal disease (ESRD) patients.[1, 2] Ertapenem is an antibiotic used for the treatment of infections caused by several organisms, including both Gram positive and negative infections.3 Although ertapenem pharmacokinetic (PK) parameters have been described in the general population, this same information for patients on peritoneal dialysis is not available.

Determining optimal antibiotic dosing recommendations for ertapenem is imperative to the health of CAPD patients in order to prevent either excess medication or sub-therapeutic doses of the drug. This study will provide clinicians with the necessary information to safely and effectively treat CAPD patients with ertapenem.

OBJECTIVE The objective of this study is to characterize the pharmacokinetic profile of ertapenem during continuous ambulatory peritoneal dialysis (CAPD).

RESEARCH DESIGN & METHODS:

Study Location This study will be conducted at an outpatient dialysis clinic (Hortense and Louis Rubin Dialysis Center, Clifton Park, NY), where all blood, dialysate, and urine sampling will occur.

Study Population To accomplish the study objective, a prospective, open-label, pharmacokinetic study of ertapenem in 8 patients on CAPD will be conducted. The desired composition of the study population will consist of approximately 4 males and 4 females, 6 of whom will be Caucasian, and 2 non-Caucasian patients. This patient composition was selected because it reflects the demographic at the Hortense and Louis Rubin Dialysis Center, Clifton Park, NY.

i. Inclusion criteria Adult patients (≥ 18 years), non-infected (afebrile, lack of constitutional symptoms and no leukocytosis), on a stable PD regimen (at least one month) are eligible for participation. Both patients with and without residual renal function will be studied. Non-anuric patients concurrently receiving medications with the potential to inhibit active tubular secretion will be allowed to enter the study after a 2-week washout period. These medications include H2-antagonists, trimethoprim, or probenecid. The patient and their physician at the Hortense and Louis Rubin Dialysis Center will contacted if any medication needs to be discontinued.

ii. Exclusion criteria Patients will be ineligible for the study if they have had peritonitis within the previous 4 weeks, clinical signs or symptoms of active infection, elevated white blood cell count, or treatment with any antibiotic within the previous 2 weeks. Patients with a hemoglobin (hgb) < 11 g/dL will be ineligible for study inclusion. Patients with stated or documented allergies to beta-lactams medications will not be eligible. Pregnant or breastfeeding women will not be eligible for inclusion. All women of child-bearing age will need to yield a serum hCG ≤ 5 mIU/mL within 2 weeks of the scheduled study day. Patients taking valproic acid will also be excluded.

Research Plan Prior to the initiation of the study protocol, informed consent will be obtained from each participant. A translator will be consulted to accommodate non-English speaking study patients.

i. Dialysis Prescription Eligible patients will receive a standardized CAPD prescription of 4 daily exchanges with 2 L of 2.5% dextrose dialysate, having dwell periods of 6 hours, 4 hours, 6 hours and 8 hours, respectively, starting 7 days prior to ertapenem administration day. On the study day, patients will perform 2 exchanges at the Hortense and Louis Rubin Dialysis Center.

ii. Pre-Ertapenem Administration Procedure Two weeks prior to the study day, all women of child-bearing age will be required to yield a negative pregnancy test (hCG ≤ 5 mIU/mL).

One week prior to the study day, a complete blood count (CBC) will be checked to ensure that the Hb concentration is ≥11 g/dL and white blood cell (WBC) count is normal (5-10,000 cells/mm3). The patients' weights will also be recorded at this time.

On the study day, patients will arrive at the dialysis clinic, drain their peritoneal cavity and instill fresh dialysate by way of the PD catheter over 5 - 10 minutes using a Y-type administration set. Spent dialysate from the preceding exchange will be drained immediately prior to the intravenous injection of ertapenem. Patients with residual renal function will urinate immediately prior to administration of ertapenem. An aliquot (10 mL) of urine will be saved and tested to ensure that no interfering substances are present that would invalidate the assay used for ertapenem determination in the urine.

Patients will have two peripheral venous catheters placed: 1) for drug administration and 2) for blood sampling purposes.

iii. Ertapenem Administration On the study day, subjects will be given ertapenem 500 mg IV over a 30 minute infusion.

iv. Blood and Dialysate Sampling Patients will perform 2 CAPD exchanges during the study period, during which 13 blood samples and 13 dialysate samples will be collected (see figure).

v. Urine Collection Non-anuric patients will be required to collect their urine during the course of the study period.

vi. Sample preparation and assay methods The urine, plasma, and dialysate concentrations of ertapenem will be determined by a high pressure liquid chromatography (HPLC) or a liquid chromatography / mass spectrometry (LCMS) device. Blood samples will be collected in standard blood collection tubes containing sodium heparin having a maximum volume of 4 mL. Samples will be stored on ice until the plasma is harvested (within 2 hours). Plasma will be obtained by placing the blood samples in a centrifuge at room temperature at approximately 3000 - 4000 rpm for 15 minutes. The plasma will then be withdrawn, split into 2 aliquots of equal volume, and transferred into separate polypropylene tubes (Tube 1, Tube 2). The tubes are pre-labeled as either Set A (Tube 1) or Set B (Tube 2). The labels will be in indelible ink. The following information will be included on the labels: sample type (plasma), dose number after which the sample was collected (i.e., dose #3), protocol number, subject number, date and time of sampling.

Similarly the dialysate and urine samples will be split into two batches and stored at -20oC until assayed. The dialysate will be mixed thoroughly. The total sample volume will be recorded. Two milliliters of dialysate will be transferred into each of the polypropylene tubes (Tube 1 and Tube 2). The tubes are pre-labeled as either Set A (Tube 1) or Set B (Tube 2). The labels will be in indelible ink. The following information will be included on the labels: sample type (dialysate), dose number after which the sample was collected (i.e., dose #3), protocol number, subject number, date and time of sampling. Samples will be stored frozen at -20 degrees Centigrade until they are shipped for concentration determination. Blank dialysate (without ertapenem in it) will also be sent for assay to assess for potential interfering substances in the assay and to serve as analytical controls for the assay. The blank dialysate samples will be 10-20 mL stored in individual polypropylene tubes, clearly marked, "dialysis blank." On a separate piece of paper, the specific concentration of each component of the dialysate fluid (i.e., electrolytes, dextrose, saline, etc.) will be included in the shipment.

Urine will be collected and split into two aliquots of equal volume and transferred to polypropylene tubes (Tube 1 and Tube 2). The tubes will pre-labeled as Tube A (Tube 1) and Tube B (Tube 2). Tubes will be pre-labeled with indelible ink and include the following information: sample type (urine), protocol number, and subject number. Samples will be stored frozen at -20 degrees Centigrade until they are shipped for ertapenem concentration determination.

One batch of dialysate samples will be packed on dry ice (sufficient for 2 days) and shipped to a location to be determined by Merck. One batch of blood and urine samples will be packed in dry ice (sufficient for 2 days) and shipped to a location to be determined by Merck. The second batch of samples (dialysate, blood, and urine) will be sent to a central laboratory (Quest Diagnostics, Inc) for serum, urine, and dialysate creatinine and urea assay and dialysate dextrose concentration assay.

Data Analysis:

All pharmacokinetic data will be analyzed in a population pharmacokinetic model using the Non Parametric Adaptive Grid with adaptive γ (NPAG) program of Leary, Schumitzky and Jelliffe.5 Upon obtaining model convergence, the mean parameter vector and covariance matrix from the population pharmacokinetic analysis will be embedded in Subroutine Prior of the ADAPT II package of programs of D'Argenio and Schumitzky.6

The following differential equations were used to characterize the PK profile of ertapenem:

〖dX〗_1/dt=R_1-(k_12+CL/V+k_13 R_2+k_13 R_3 ) X_1+k_21 X_2+k_31 X_3 R_2+k_31 X_4 R_3 〖dX〗_2/dt=k_12 X_1-k_21 X_2 〖dX〗_3/dt=k_13 X_1 R_2-k_31 X_3 R_2 〖dX〗_4/dt=k_13 X_1 R_3-k_31 X_4 R_3+R_4 R_5 〖CONEX〗_1

where X1: amount of drug in the central compartment; X2: amount of drug in the peripheral compartment; X3: amount of drug in the first peritoneal exchange; X4: amount of drug in the second peritoneal exchange; CL: non-dialytic clearance from central compartment (liters per hour); V: volume of the central compartment (liters); k12 and k21: first-order intercompartmental transfer rate constants between central and peripheral compartments (inverse hours); k13 and k31: first-order intercompartmental transfer rate constants between central and peritoneal compartments; CONEX1: amount of ertapenem remaining in peritoneal compartment after drainage of first study exchange (mg); R1: time-delimited zero-order drug input rate (piece-wise input function) into central compartment (mg per hour); R2: rate constant for first dwell constrained to 0 (first dwell turned off) or 1 (first dwell turned on); R3: rate constant for second dwell constrained to 0 (second dwell turned off) or 1 (second dwell turned on); R4: ertapenem dialysate concentration observed at the end of the first dwell; R5:input rate for residual amount of dialysate volume remaining after drainage of the first dwell.

The population simulation without process noise option will be employed. A 9,999 subject Monte Carlo simulation will be performed to examine an array of potential ertapenem candidate dosing regimens in CAPD.

REFERENCES

1. Bloembergen WE, Port FK. Epidemiological perspective on infections in chronic dialysis patients. Adv Ren Replace Ther. Jul 1996;3(3):201-207.
2. United States Renal Data System. USRDS Annual Data Report: Atlas of End-stage Renal Disease in the United States. Bethesda, MD: National Institute of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2007.
3. Merck & Co, Inc. Invanz (ertapenem) package insert. Whitehouse Station, NJ; 2008.
4. D'Argenio DZ, Schumitzky A. A program package for simulation and parameter estimation in pharmacokinetic systems. Comput Programs Biomed. Mar 1979;9(2):115-134.
5. Leary, R., R. Jelliffe, A. Schumitzky, and M. van Guilder. An adaptive grid, non-parametric approach to pharmacokinetic and dynamic (PK/PD) models. Proceedings, Fourteenth IEEE Symposium on Computer-Based Medical Systems. 26-27 July 2001. Bethesda, MD, IEEE Computer Society, pp. 389-394.
6. D'Argenio, D. Z., and A. Schumitzky. 1979. A program package for simulation and parameter estimation in pharmacokinetic systems. Comput Programs Biomed 9:115-34.

ELIGIBILITY:
i. Inclusion criteria Adult patients (≥ 18 years), non-infected (afebrile, lack of constitutional symptoms and no leukocytosis), on a stable PD regimen (at least one month) are eligible for participation. Both patients with and without residual renal function will be studied. Non-anuric patients concurrently receiving medications with the potential to inhibit active tubular secretion will be allowed to enter the study after a 2-week washout period. These medications include H2-antagonists, trimethoprim, or probenecid. The patient and their physician at the Hortense and Louis Rubin Dialysis Center will contacted if any medication needs to be discontinued.

ii. Exclusion criteria Patients will be ineligible for the study if they have had peritonitis within the previous 4 weeks, clinical signs or symptoms of active infection, elevated white blood cell count, or treatment with any antibiotic within the previous 2 weeks. Patients with a hemoglobin (hgb) < 11 g/dL will be ineligible for study inclusion. Patients with stated or documented allergies to beta-lactams medications will not be eligible. Pregnant or breastfeeding women will not be eligible for inclusion. All women of child-bearing age will need to yield a serum hCG ≤ 5 mIU/mL within 2 weeks of the scheduled study day. Patients taking valproic acid will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie E Cardone, PharmD, Principal Investigator — Albany College of Pharmacy and Health Sciences
Locations (1):
- Hortense and Louis Rubin Dialysis Center, Clifton Park, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from an outpatient dialysis center. Eligible patients were referred to study investigators by social workers or nurses.
Pre-assignment Details: All study patients were assigned to receive study drug to explore the pharmacokinetic profile of ertapenem during CAPD. Once enrolled, patients were excluded if they developed infection.
Period: Overall Study
Arm/Group | Ertapenem 500 mg IV x1
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 55.14 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Volume of Distribution, Central Compartment (Vc)
Description: Population PK
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
Liters (L) | 2.78 (062)

2. Primary Outcome: Clearance (CL)
Description: population PK clearance
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: Liters/hour (L/h)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
Liters/hour (L/h) | .24 (.068)

3. Primary Outcome: k12
Description: 1st order intercompartmental rate constant between central and peripheral compartments
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: h^(-1)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
h^(-1) | 2.51 (1.39)

4. Primary Outcome: k21
Description: 1st order intercompartmental rate constant from peripheral to central compartment
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: h^(-1)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
h^(-1) | 2.03 (1.04)

5. Primary Outcome: k13
Description: 1st order intercompartmental rate constant from central to peritoneal cavity
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: h^(-1)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
h^(-1) | 0.082 (.053)

6. Primary Outcome: k31
Description: 1st order intercompartmental rate constant peritoneal cavity to central
Time Frame: 12h
Measure: Mean (Standard Deviation); unit: h^(-1)
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
h^(-1) | .16 (.074)

7. Primary Outcome: Residual Drug in Peritoneal Cavity After 1st Exchange
Time Frame: 6h
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ertapenem 500 mg IV x1
Number analyzed (Participants) | 7
mg | .64 (.43)

ADVERSE EVENTS:
Arm/Group | Ertapenem 500 mg IV x1
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less